CLINICAL TRIAL: NCT03621371
Title: Metacognitive Therapy and Intolerance of Uncertainty Therapy for Generalized Anxiety Disorder in Primary Care: Randomized Controlled Pilot Study
Brief Title: Cognitive-behavioral Therapy for Generalized Anxiety Disorder in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Benjamin Bohman, Dr, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLSO-2018/505-31/1
Record Dates: First submitted 2018-06-28; First posted 2018-08-08 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metacognitive therapy (Experimental)
  Interventions: Behavioral: Metacognitive therapy
- Intolerance of uncertainty therapy (Experimental)
  Interventions: Behavioral: Intolerance of uncertainty therapy

INTERVENTIONS:
Behavioral: Metacognitive therapy — Metacognitive therapy is a form av cognitive-behavioral therapy which aims to change cognitions about worry in patients with generalized anxiety disorder.
  Arms: Metacognitive therapy
Behavioral: Intolerance of uncertainty therapy — Intolerance of uncertainty therapy is a form av cognitive-behavioral therapy which aims to reduce cognitive and behavioral avoidance of uncertain situations or cognitions which lead to worry in patients with generalized anxiety disorder.
  Arms: Intolerance of uncertainty therapy

SUMMARY:
The feasibilty and preliminary comparative effectiveness of two methods of cognitive-behavioral therapy - metacognitive therapy and intolerance of uncertainty therapy - for primary care patients with generalized anxiety disorder is investigated in a pilot study using a randomized controlled design. Purpose of the study is to examine the feasibility of a full-scale randomized controlled trial. Research questions primarily concern recruitment, measurement, and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of generalized anxiety disorder
* Age 18 years or above
* Being able to understand and speak Swedish without interpreter support

Exclusion Criteria:

* Psychosis, bipolar disorder, severe depressive symptoms, risk of suicid, substance use disorder, intellectual disability
* Simultaneous psychological treatment
* If pharmacological treatment, it needs to be stable prior to and during treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Liljeholmen Primary Health Care Center, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Af Winklerfelt Hammarberg S, Toth-Pal E, Jansson-Frojmark M, Lundgren T, Westman J, Bohman B. Intolerance-of-uncertainty therapy versus metacognitive therapy for generalized anxiety disorder in primary health care: A randomized controlled pilot trial. PLoS One. 2023 Jun 14;18(6):e0287171. doi: 10.1371/journal.pone.0287171. eCollection 2023. PMID 37315099

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metacognitive Therapy | Intolerance of Uncertainty Therapy
Started | 31 | 33
Completed | 25 | 32
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metacognitive Therapy | Intolerance of Uncertainty Therapy | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.8) | 37.1 (11.6) | 36.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Penn State Worry Questionnaire - Measure of Symptom Change
Description: Penn State Worry Questionnaire, a self-reported symptom measure of worry. Scale ranges: 16-80 scores on a scale; higher values represent a worse outcome.
Time Frame: Change from baseline symptoms at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metacognitive Therapy | Intolerance of Uncertainty Therapy
Number analyzed (Participants) | 31 | 33
score on a scale | 42.1 (7.5) | 55.8 (7.5)
Statistical Analysis 1: Comparison: Metacognitive Therapy vs Intolerance of Uncertainty Therapy; Test type: Other; p < 0.05, Mixed Models Analysis; F-test = 9.88

ADVERSE EVENTS:
Time Frame: Not assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not assessed.
Arm/Group | Metacognitive Therapy | Intolerance of Uncertainty Therapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT03621371/Prot_SAP_000.pdf